CLINICAL TRIAL: NCT04778020
Title: International COVID-19 Clinical Evaluation Registry -2 (HOPE-2)
Acronym: HOPE-2
Status: Completed | Type: Observational
Sponsor: St Carlos Hospital, Madrid, Spain (Other)
Responsible Party: Principal Investigator, IVAN J NUÑEZ GIL, MD, PhD, MSc. Principal Investigator, St Carlos Hospital, Madrid, Spain
Other Study IDs: 21/128-E
Record Dates: First submitted 2021-02-20; First posted 2021-03-02 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PURPOSE. The main objective of the present study is to carefully characterize the clinical profile of individuals with lasting sequelae after a COVID-19 admission.

As secondary objectives, the analysis of the risk-adjusted influence of COVID-19 severity, previous comorbidities and management of patients discharged after COVID-19 will be performed.

DESIGN AND STATISTICAL ANALYSIS Cross-sectional and prospective registry, a real life "all comers" type, with voluntary participation, without specific funding or conflicts of interest.

It is a study initiated by researcher that will have advanced statistical support from the IMAS foundation (Institute for the Improvement of Health Care, Madrid, Spain) and the Cardiovascular Research Foundation (FIC, Madrid, Spain).

International level.

PARTICIPANTS PROTOCOL. The study has been approved by Hospital Clinico San Carlos Ethic´s Committee (21/128-E) and the institutional board of each participating center.

The present study proposes the continuation in time of the work previously carried out in the HOPE registry.

It proposes to select all the patients attended in any health center (with in hospital beds), who have been discharged or have died up to 31st august 2020.

All will be considered eligible with a positive COVID-19 test (any type) or if their attending physicians consider them highly likely to have presented the infection.

Given the anonymous characteristics of the registry and the health alarm situation generated by the virus, in principle, it is not considered necessary to provide written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged (deceased or alive) from any hospital center with a confirmed diagnosis.

Exclusion Criteria:

* There are no exclusion criteria, except for the patient's explicit refusal to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Same inclusion/exclusion as HOPE COVID-19. We propose the long-term follow-up of patients discharged after a COVID-19 admission up to 31st august 2020.
  Consecutive inclusion and the completion of patients previously included in HOPE registry is strongly warranted.
Sampling Method: Non-Probability Sample
Enrollment: 9299 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
DEATH | through study completion, an average of 1 year
  Number of participants dead by any cause during follow up.

SECONDARY OUTCOMES:
Any POSTCOVID-19 symptom | through study completion, an average of 1 year
  Events defined in HOPE 2 protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study termination